CLINICAL TRIAL: NCT03698461
Title: Comparative Analysis of Immune Profile Following Neoadjuvant Chemotherapy in Colorectal Liver Metastases (CRLM): A Prospective Pilot Clinical Trial
Brief Title: Treatment of Colorectal Liver Metastases With Immunotherapy and Bevacizumab
Acronym: CLIMB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Sun Young Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASA-1
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — atezolizumab; Bevacizumab; Oxaliplatin; Levoleucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab, Bevacizumab, FOLFOX (Experimental): Atezolizumab 1200mg IV Once, Atezolizumab (840mg IV D1 of C1-12) + Bevacizumab (5mg/kg IV D1 of C1-12) + FOLFOX(Oxaliplatin 85mg/m2 IV D1 of C1-12, Levoleucovorin 200mg/m2 IV D1 of C1-12, 5-FU - bolus 400mg/m2 IV D1 of C1-12, - infusional 2400mg/m2 IV continuous(46 hours) D1-3 of C1-12)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Levoleucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: Atezolizumab — * 1200mg IV on day1 before start of cycle 'atezolizuamb, bevacizumab + FOLFOX(Oxaliplatin, Levoleucovorin, 5-FU')
  * 840mg IV D1 of C1-12 (Cycle: every 2 weeks)
  Other Names: Tecentriq
Drug: Bevacizumab — 5mg/kg IV D1 of C1-12 (Cycle: every 2 weeks) at least 5 minutes after completion of atezolizumab
  Other Names: Avastin
Drug: Oxaliplatin — 85mg/m2 IV D1 of C1-12 (Cycle: every 2 weeks)
Drug: Levoleucovorin — 200mg/m2 IV D1 of C1-12 (Cycle: every 2 weeks)
Drug: 5-FU — * 5-FU Bolus: 400mg/m2 IV bolus D1 of C1-12 (Cycle: every 2 weeks)
  * 5-FU infusion: 2400mg/mg continuous IV infusion over 46hours D1-3 of C1-12 (Cycle: every 2 weeks)
  Other Names: 5-fluorouracil

SUMMARY:
Liver is the most common site of metastases from colorectal cancer. Neoadjuvant chemotherapy with targeted agents is usually recommended for borderline-resectable liver metastases that are technically difficult to resect for conversion to resectable disease and control of metastatic spread. However, the prognosis of these patients are still poor, and long term disease-free survival over 3 years is rare and <20%. More effective measures to prevent recurrence are needed before or after resection of colorectal liver metastases.

DETAILED DESCRIPTION:
* Atezolizumab is a humanized immunoglobulin G1 monoclonal antibody that targets Programmed Death-Ligand 1(PD-L1) and inhibits the interaction between PD-L1 and its receptors, Programmed cell Death protein 1(PD-1) and B7.1. Therapeutic blockade of PD-L1 binding by atezolizumab has been shown to enhance the magnitude and quality of tumor specific T cell responses, resulting in improved anti tumor activity.
* Bevacizumab is a recombinant, humanized therapeutic antibody directed against vascular endothelial growth factor(VEGF). In addition to its well-characterized role in angiogenesis, VEGF is also believed to be involved in cancer immune evasion via the induction of myeloid- derived suppressor cells(MDSCs). These VEGF-induced MDSCs can suppress both T-cell and dendritic-cell function. Bevacizumab can restore and/or maintain the antigen presentation capacity of dendritic cells, leading to enhanced T-cell infiltration in tumors. When used in combination, VEGF targeting agents such as bevacizumab promote the normalization of tumor vasculature and may thereby increase access of therapeutic agents.
* Atezolizumab with bevacizumab, levoleucovorin, oxaliplatin, and 5-fluorouracil(FOLFOX). A translational study for renal cell carcinoma showed bevacizumab resulted in modulation of tumor immune microenvironment with Th1-related signatures, which was more potentiated by subsequent treatment with atezolizumab. This suggests potentiation of anti-tumor immunity with the combination of bevacizumab and atezolizumab.

ELIGIBILITY:
<Inclusion Criteria>

Patient-related consideration

1. Have provided written informed consent prior to any study specific procedures
2. Willing and able to comply with the protocol
3. ≧ 20 years of age at the time of signing Informed Consent Form
4. Eastern Cooperative Oncology Group (ECOG) status of ≤1

Disease-related consideration

1. Histologically diagnosed colorectal adenocarcinoma
2. Liver metastases from colorectal adenocarcinoma confirmed through biopsy
3. Liver metastatic lesions should be considered to be potentially resectable after conversion chemotherapy by multi-disciplinary team and should meet one of the following criteria:

   * Number of metastatic deposit ≧ 4
   * Possibility of resection margin could be involved
   * Involvement of major hepatic vessels
   * Presence of extrahepatic metastases (if they are supposed to be treated with curative aim and not to alter a plan for hepatic metastasectomy)
   * High likelihood of insufficient residual hepatic volume after surgery
4. Measurable by RECIST criteria 1.1.
5. One or more hepatic lesions should be accessible for biopsy
6. Archival tumor tissue from the metastatic liver lesion obtained at the time of the initial diagnosis must be available.
7. Adequate major organ functions as following:

   * Hematopoietic function: Absolute neutrophil count(ANC) ≧ 1,500/mm3, Platelet ≧ 100,000/mm3
   * Hepatic function: serum bilirubin ≦ 2 x Upper limit of normal(ULN), Aspartate aminotransferase(AST)/Alanine aminotransferase(ALT) ≦ levels 5 x ULN
   * Renal function: serum creatinine ≦ 1.5 x ULN
8. International normalised ratio(INR) < 1.5 or Activated partial thromboplastin(aPTT) < 1.5 x ULN within 14 days prior to the start of study treatment for patients not receiving anti-coagulation. For patients receiving anticoagulants, INR and aPTT must be within the medical standard of enrolling institution.

Other considerations

1. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment after the last dose of study treatment

   i. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≧12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

   ii. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
2. For men, they must practice abstinence or condom use, and abstain from sperm donation during the treatment period and for 6 months after their last dose of study treatment during the treatment period and for 6months after the last dose of study treatment.

<Exclusion Criteria>

Patients who meet any of the following criteria will be excluded from study entry:

1. Extrahepatic metastases that are not candidates for treatment of curative aim (e.g. resection, radiation or radiofrequency ablation)
2. Presence of central nervous system (CNS) metastases
3. Concurrent or previous history of another primary cancer within 3 years prior to study treatment except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis or pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the principal investigator.
4. Chronic alcoholic hepatitis or cirrhosis
5. Chronic hepatitis B, defined as HBV DNA (> 2,000 IU / mL) and ALT> upper limit of normal range, must be treated with antiviral drugs before enrollment to reach appropriate viral suppression (HBV DNA <2000 IU / mL), and the antiviral drugs must be maintained during the study treatment period and for 6 months after the last dose of study treatment.
6. Prior chemotherapy for metastatic disease
7. Uncontrolled medical illness congestive heart failure, myocardial infarction within 6 months including medically uncontrolled infection, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months
8. Prior adjuvant FOLFOX chemotherapy
9. Prior adjuvant chemotherapy, if administered within 6 months before study entry
10. Current or recent (within 10 days of start of study treatment) use of aspirin (>325mg/day), clopidogrel (>75mg/day), therapeutic or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (therapeutic anticoagulation on a stable dose for at least 2 weeks prior to the start of study treatment is allowed)
11. Known alcohol or drug abuse
12. Active infection requiring intravenous antibiotics at the start of study treatment
13. Inadequately controlled hypertension (defined as systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg)
14. Prior history of hypertensive crisis or hypertensive encephalopathy
15. History or evidence upon physical or neurological examination of CNS disease (e.g. seizures) unrelated to cancer unless adequately treated with standard medical therapy
16. Uncontrolled chronic peripheral neuropathy ≥ CTCAE grade 2
17. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of start of study treatment
18. Any previous venous thromboembolism > CTCAE Grade 3 within 12 months prior to start of study treatment
19. History of haemoptysis ≥ Grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month of start of study treatment
20. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation)
21. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to start of study treatment, or anticipation of need for major surgical procedure (other than hepatic metastasectomy) during the course of the study
22. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to start of study treatment
23. Serious, non-healing wound, active ulcer, or untreated bone fracture
24. Known hypersensitivity to any component of any of the study medication
25. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins
26. Known dihydropyrimidine dehydrogenase deficiency
27. Pregnant or breastfeeding, or intending to become pregnant during the study or within 6 months after the last dose of study treatment
28. Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to initiation of study treatment.
29. Known hypersensitivity or allergy to Chinese hamster ovary cell products
30. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      * Rash must cover 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
31. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
32. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted.)
33. Positive test for human immunodeficiency virus (HIV)
34. Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening

    * The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
    * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
35. Active tuberculosis
36. Administration of a live, attenuated vaccine within 4 weeks prior to start of study maintenance treatment or anticipation that such a live attenuated vaccine will be required during the study
37. Prior treatment with Cluster of differentiation(CD)137 agonists, anti-cytotoxic T-lymphocyte-associated antigen(CTLA)4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
38. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of study maintenance treatment
39. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-Tumour Necrosis Factor agents) within 2 weeks prior to start of study maintenance treatment, or requirement for systemic immunosuppressive medications during the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Serial changes in Cluster of Differentiation(CD) 8+ T cell densities | Baseline, Day15 of first atezolizumab administration, and after at least 6 cycles (each cycle is 14days)
  Opal(TM) platform Immunohistochemistry(IHC)

SECONDARY OUTCOMES:
Serial changes of Immune cell biomarkers CD3, CD4, Programmed death-Ligand 1(PD-L1),PD-1, granzyme B, CD45RO, Forkhead Box P3(FOXP3), CD68 | Baseline, Day15 of atezolizumab, and after at least 6 cycles (each cycle is 14days)
  Opal(TM) platform IHC
Serial changes of Immune cell CD3+, CD8+ densities | Baseline, Day15 of atezolizumab, and after at least 6 cycles (each cycle is 14days)
  IMMUNOSCORE® (IMMUNOSCORE is a registered trademark owned by INSERM)
Serial changes of Density of Vascular marker CD31, CD34 | Baseline, Day15 of atezolizumab, and after at least 6 cycles (each cycle is 14days)
  Opal(TM) platform IHC
Serial changes of Gene expression profile | Baseline, Day15 of atezolizumab, and after at least 6 cycles (each cycle is 14days)
  RNA-seq
Response Rate | Baseline, at 6th week from the first treatment, and then every 6±2 weeks up to 12 cycles (each cycle is 14days), every 3 months after the 12 cycles up to 24months
  RECIST 1.1 and immune RECIST(iRECIST)
Progression-Free Survival | Baseline, at 6th week from the first treatment, and then every 6±2 weeks up to 12 cycles (each cycle is 14days), every 3 months after the 12 cycles up to 24months
  RECIST 1.1 and iRECIST
R0 resection rate | At the time of hepatic resection
  All gross lesions are resected and all surgical margins are free from tumor cells (The proportion of patients who undergo R0 resection for liver metastases out of all patients who started at least one dose of study treatment.)
Incidence, nature and severity of adverse events with severity (Safety profile) | Consent to 90 days after the last dose of investigational medicinal product or until initiation of new systemic anti-cancer therapy, whichever occurs first.
  Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Microbiome profile | Day1 before first atezolizumab administration, Day15 before the treatment and at time of hepatic metastasectomy or liver biopsy after 6 cycles of treatment (each cycle is 14days)
  In stool samples through whole metagenomic sequencing

CONTACTS AND LOCATIONS:
Overall Officials: SunYoung Kim, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No